CLINICAL TRIAL: NCT05541146
Title: Evaluation of Intraperitoneal Chemotherapy in the Treatment of Gastric Cancer in Patients With Peritoneal Carcinomatosis
Brief Title: Intraperitoneal Chemotherapy in Gastric Cancer With Peritoneal Carcinomatosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP 1507/19; 26306419.8.0000.0065 (Registry Identifier: Plataforma Brasil - CAAE); 2020/13249-0 (Other Grant/Funding Number: The Sao Paulo Research Foundation, FAPESP)
Record Dates: First submitted 2022-08-23; First posted 2022-09-15 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2022-09

CONDITIONS: Gastric Cancer; Peritoneal Carcinomatosis
Keywords: Gastric Cancer; intraperitoneal chemotherapy; gastric adenocarcinoma; conversion surgery; stage IV gastric cancer; peritoneal metastases; carcinomatosis
MeSH Terms: conditions — Stomach Neoplasms; Peritoneal Neoplasms; Carcinoma | interventions — Hyperthermic Intraperitoneal Chemotherapy; Drug Therapy; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Patients will undergo intraperitoneal chemotherapy with Paclitaxel (4 cycles) associated with systemic chemotherapy. After treatment, patients will be reassessed and if there is a peritoneal response, they will undergo gastrectomy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intraperitoneal chemotherapy (Experimental): Intraperitoneal chemotherapy in gastric cancer patients with peritoneal carcinomatosis.
  Interventions: Combination Product: Intraperitoneal chemotherapy

INTERVENTIONS:
Combination Product: Intraperitoneal chemotherapy — Patients will undergo intraperitoneal chemotherapy with Paclitaxel (4 cycles) associated with systemic chemotherapy. After treatment, patients will be reassessed and if there is a peritoneal response, they will undergo gastrectomy
  Other Names: Implantation of intraperitoneal catheter for chemotherapy with Paclitaxel

SUMMARY:
Peritoneal carcinomatosis (PC) in gastric cancer (GC) is considered a fatal disease, without expectation of definitive cure. Since conventional surgery is not indicated in the palliative setting, and systemic chemotherapy treatments are not sufficient to contain the disease, a multimodal approach associating intraperitoneal (IP) chemotherapy (CMT) with surgery may represent an alternative for these patients.

IP CMT has shown superior results to conventional treatment in patients at this stage of the disease, and can achieve complete regression of lesions in a significant portion of cases. Once response to treatment is achieved, patients become fit for curative surgery, which offers a new perspective on the survival in these previously unresectable cases, and raising survival rates to similar levels to patients undergoing surgery with curative intention.

Thus, the aim of this study is to evaluate the complete response rate and curative resection in patients with PC by GC at Instituto do Cancer do Estado de São Paulo (ICESP) treated with IP CMT. Patients prospectively included in the study will undergo implantation of a peritoneum catheter to perform outpatient IP CMT in order to promote the regression of lesions. Those with complete regression may be referred for surgical treatment, curing a portion of these patients. The diagnosis of PC will be performed by conventional cytological, immunohistochemical and liquid cytology methods to determine the presence of tumor cells in the peritoneal lavage and to evaluate the sensitivity of the methods. In addition, it is proposed in the study the storage of material for further study of circulating markers in peripheral blood and peritoneal lavage that may be related to response or resistance to treatment.

It is believed that IP CMT may not only increase the survival of patients with PC, but also offer the possibility of cure for a significant portion of patients who are currently without treatment prospects and with a median survival of only six months.

DETAILED DESCRIPTION:
This is a prospective study lasting 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Gastric adenocarcinoma
* Presence of peritoneal carcinomatosis documented through intraoperative identification and confirmed by biopsies and/or positive oncotic cytology;
* Presence of exclusively peritoneal metastasis with PCI < 12;
* Age between 18 and 75 years;
* Eastern Cooperative Oncology Group (ECOG) performance scale 0 and 1;
* Body mass index (BMI) greater than 18;
* Total WBC count ≥3000, neutrophils ≥1500, hemoglobin ≥8, and platelet count ≥100,000;
* Bilirubin <2, TGO/TGP/FA/GGT 3x the reference value;
* Creatinine clearance calculated by the Cockcroft-Gault formula ≥ 50 ml/min.

Exclusion Criteria:

* Synchronous or metachronic neoplasms;
* Previous antineoplastic treatment for gastric cancer;
* Clinical conditions considered critical by the investigator;
* Obstruction of the digestive tract;
* Suspected gastrointestinal bleeding;
* New York Heart Association functional class II/III/IV heart failure;
* Heart disease that, in the opinion of the investigator, prevents the patient from receiving the necessary hydration during chemotherapy with cisplatin.
* Known HIV infection or chronic use of immunosuppressants;
* Acute myocardial infarction or stroke in the last 6 months
* pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Rate of complete peritoneal response after 04 cycles of intraperitoneal (IP) chemotherapy (CMT) associated with systemic CMT with XP. | At the end of Cycle 4 (each cycle is 8 days)
  Absence of visible carcinomatosis on imaging tests, absence of viable peritoneal lesion at laparoscopy and absence of neoplastic cells in peritoneal lavage.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 6 months
  Time between conversion surgery and date of disease progression, assessed in the first 6 months
Overall survival (OS) | 5 years
  Time between conversion surgery and last follow-up after 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Andre Roncon Dias, MD, PhD, Principal Investigator — Instituto do Câncer de São Paulo - ICESP
Locations (1):
- Instituto do Câncer de São Paulo - ICESP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No